CLINICAL TRIAL: NCT07362654
Title: Single-cell Study of the Systemic Immune Response to Controlled Gluten Intake in Pediatric Celiac Disease
Brief Title: Single-cell Immune Response to Controlled Gluten Ingestion in Pediatric Celiac Disease
Acronym: CELLiomicS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Collaborators: Hospital Regional de Malaga (Other); Andaluz Health Service (Other Government); Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental (Other); Universidad de Málaga (Unknown); Centro de Investigación Biomédica (Unknown); Biohealth Research Institute in Granada (ibs.GRANADA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PI-0070-2024
Record Dates: First submitted 2025-12-17; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-11

CONDITIONS: Celiac Disease; Gluten Sensitivity; Autoimmune Diseases
Keywords: Celiac Disease; Gluten Exposure; Single-Cell RNA Sequencing; Gluten-Free Diet; Immune Response; Pediatrics; Omics
MeSH Terms: conditions — Celiac Disease; Autoimmune Diseases | interventions — Glutens; Defecation

STUDY DESIGN:
Intervention Model Description: Participants with celiac disease are randomized into three parallel intervention groups receiving placebo, 50 mg gluten, or 5 g gluten.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple-blind (participant, care provider, investigator, outcomes assessor). Only three designated team members not involved in routine clinical assessment or outcome evaluation have access to the randomization list in order to prepare the gluten/placebo doses and monitor safety. Data entry and statistical analyses are performed using a blinded database.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo Group (Placebo Comparator): Participants receive a placebo preparation once daily on Days 1, 2, and 3. Blood samples are collected on Day 1 (baseline) and Day 8 (post-intervention). Participants and evaluators remain blinded to allocation.
  Interventions: Dietary Supplement: Placebo; Procedure: Collection of blood, stool and urine samples on Day 1 and Day 8.
- Low-Dose Gluten (50 mg) (Experimental): Participants receive 50 mg of gluten once daily on Days 1, 2, and 3, simulating accidental low-level exposure. Blood samples are collected on Day 1 (baseline) and Day 8 (post-intervention). Participants and evaluators remain blinded to allocation.
  Interventions: Dietary Supplement: Gluten 50 mg; Procedure: Collection of blood, stool and urine samples on Day 1 and Day 8.
- High-Dose Gluten (5 g) (Experimental): Participants receive 5 g of gluten once daily on Days 1, 2, and 3, simulating a dietary transgression. Blood samples are collected on Day 1 (baseline) and Day 8 (post-intervention). Participants and evaluators remain blinded to allocation.
  Interventions: Dietary Supplement: Gluten 5 g; Procedure: Collection of blood, stool and urine samples on Day 1 and Day 8.

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo preparation identical in appearance and administration schedule to gluten doses. Administered once daily on Days 1, 2, and 3. Used as the comparator. Participants and evaluators remain blinded to allocation.
  Arms: Placebo Group
Dietary Supplement: Gluten 50 mg — Participants receive 50 mg of gluten once daily on Days 1, 2, and 3. This dose simulates accidental low-level gluten exposure in children with celiac disease. Participants and evaluators remain blinded to allocation.
  Arms: Low-Dose Gluten (50 mg)
Dietary Supplement: Gluten 5 g — Participants receive 5 g of gluten once daily on Days 1, 2, and 3. This dose simulates a dietary transgression in children with celiac disease. Participants and evaluators remain blinded to allocation.
  Arms: High-Dose Gluten (5 g)
Procedure: Collection of blood, stool and urine samples on Day 1 and Day 8. — In addition to blood samples, stool and urine samples will be collected for complementary analyses (including fecal gluten immunogenic peptides (GIP) and exploratory metabolomic assays)

SUMMARY:
This study investigates how the immune system of children with celiac disease responds to controlled, small amounts of gluten. Children on a strict gluten-free diet are randomly assigned to receive either placebo, 50 mg of gluten, or 5 g of gluten once daily for three days, simulating real-life accidental exposure or dietary transgression. Blood samples are collected on Day 1 (before gluten intake) and Day 8 (five days after the last dose). Stool and urine samples are also collected for complementary analyses.

Using single-cell ribonucleic acid (RNA) sequencing, T-cell receptor sequencing, microRNA profiling, and exploratory metabolomics, the study aims to characterize changes in immune cell populations and gene expression after gluten exposure. The objective is to determine whether even very small amounts of gluten induce measurable systemic immune responses and whether these responses differ according to the dose administered. Understanding these mechanisms may support the development of new biomarkers and improve clinical management of pediatric celiac disease.

DETAILED DESCRIPTION:
Celiac disease is a chronic, immune-mediated enteropathy triggered by gluten ingestion in genetically predisposed individuals. In pediatric patients, strict adherence to a gluten-free diet (GFD) leads to mucosal recovery and clinical improvement; however, the systemic immunological landscape during long-term GFD remains incompletely understood. Accidental gluten exposure is common in daily life and may trigger subclinical immune activation even in the absence of overt symptoms. The biological consequences of such low-dose exposures, particularly at the single-cell level, are not fully characterized in children.

CELLiomicS (Single-cell Immune Response to Controlled Gluten Ingestion in Pediatric Celiac Disease) is a randomized, controlled, parallel-group clinical study designed to characterize systemic immune responses to controlled gluten ingestion in pediatric patients with established celiac disease. Eligible participants are children aged 8-14 years who have followed a strict GFD for at least 18 months before enrollment. The study plans to recruit approximately 45 participants with biopsy- or serology-confirmed celiac disease.

Participants are randomized into three intervention groups: placebo, 50 mg gluten, or 5 g gluten. The selected gluten doses represent two clinically relevant scenarios: (1) accidental low-level exposure (50 mg), and (2) dietary transgression (5 g), both below the threshold typically required to cause serological relapse. Gluten or placebo is administered once daily on Days 1, 2, and 3. Blood samples are obtained on Day 1 (baseline) and Day 8 (five days after the final dose). Stool and urine samples are also collected at the same time points for complementary analyses, including fecal gluten immunogenic peptides (GIP) and exploratory metabolomics.

Peripheral blood mononuclear cells are processed for high-dimensional immune profiling using single-cell RNA sequencing and T-cell receptor (TCR) sequencing (10x Genomics). These analyses enable characterization of immune cell composition, transcriptional activity, and clonal T-cell dynamics before and after gluten challenge. In addition, exosomal microRNA expression is assessed as approved by the ethics committee amendment SICEIA-2025-001434, and untargeted metabolomic profiling of blood, stool, and urine samples is performed to explore systemic metabolic signatures associated with gluten exposure.

The primary objective is to identify gluten-induced transcriptional and cellular changes in peripheral immune cells between baseline (Day 1) and post-intervention (Day 8). Secondary objectives include: (1) assessing dose-dependent immune activation; (2) identifying immune cell subsets and gene expression programs associated with different gluten quantities; (3) characterizing TCR repertoire alterations following gluten exposure; (4) evaluating inter-individual variability in immune responses; (5) analyzing exosomal microRNA changes; and (6) identifying metabolomic signatures associated with gluten ingestion.

By providing a high-resolution view of systemic immune activation following controlled gluten ingestion, this study aims to deepen understanding of the biological impact of real-world gluten exposure in pediatric celiac disease and to support the development of novel biomarkers for dietary monitoring and personalized clinical management.

ELIGIBILITY:
Inclusion Criteria:

* Age 8 to 14 years at study entry.
* Diagnosis of celiac disease according to ESPGHAN 2020 criteria.
* At least 18 months on a strict gluten-free diet (GFD).
* Adequate adherence to the GFD, demonstrated by negative fecal gluten immunogenic peptides (GIP) prior to inclusion.
* Asymptomatic from a gastrointestinal perspective in the preceding weeks.
* Ability to swallow the gluten/placebo preparation.
* Written informed consent from parents/legal guardians and assent from the child.

Exclusion Criteria:

* Obesity defined as BMI ≥ 95th percentile according to WHO criteria.
* Diagnosed inflammatory bowel disease or diabetes mellitus.
* Acute infectious illness at the time of inclusion.
* Chronic hepatic, pulmonary, renal, or rheumatologic disease.
* History of severe acute reactions to accidental gluten ingestion.
* Use of oral corticosteroids or immunosuppressive therapy in the previous 3 months.
* Any condition that, in the opinion of the investigators, may contraindicate participation or compromise study integrity.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in peripheral blood immune cell gene expression after controlled gluten ingestion | Day 1 to Day 8
  Change from baseline (Day 1) to post-intervention (Day 8) in gene expression profiles of peripheral blood immune cells measured by single-cell RNA sequencing (scRNA-seq).
Change in peripheral blood T-cell receptor repertoire after controlled gluten ingestion | Day 1 to Day 8
  Change from baseline (Day 1) to post-intervention (Day 8) in T-cell receptor (TCR) diversity and clonality in peripheral blood T cells measured by TCR sequencing

SECONDARY OUTCOMES:
Dose-dependent changes in immune gene expression after gluten exposure | Day 1 to Day 8
  Change from baseline (Day 1) to post-intervention (Day 8) in immune-related gene expression levels measured by single-cell RNA sequencing (scRNA-seq), comparing placebo, 50 mg gluten, and 5 g gluten groups.
Dose-dependent changes in T-cell receptor repertoire clonality after gluten exposure | Day 1 to Day 8
  Change from baseline (Day 1) to post-intervention (Day 8) in T-cell receptor (TCR) clonality and diversity measured by TCR sequencing, comparing placebo, 50 mg gluten, and 5 g gluten groups.
Inter-individual variability in immune gene expression response to gluten exposure across participants | Day 1 to Day 8
  Inter-individual variability in changes from baseline (Day 1) to post-intervention (Day 8) in immune gene expression profiles measured by single-cell RNA sequencing (scRNA-seq).
Changes in serum exosomal microRNA expression after gluten exposure | Day 1 to Day 8
  Change from baseline (Day 1) to post-intervention (Day 8) in serum exosomal microRNA expression levels.
Changes in metabolomic profiles after gluten exposure | Day 1 to Day 8
  Change from baseline (Day 1) to post-intervention (Day 8) in untargeted metabolomic profiles measured in blood, stool, and urine samples.
Changes in peripheral blood immune cell type proportions after gluten exposure | Day 1 to Day 8
  Change from baseline (Day 1) to post-intervention (Day 8) in the relative proportions of immune cell types identified in peripheral blood by single-cell RNA sequencing (scRNA-seq).

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Martín Masot, MD, PhD, Principal Investigator — Hospital Regional Universitario de Málaga / IBIMA-BIONAND; Lara María Bossini Castillo, MD, PhD, Principal Investigator — IBS Granada
Locations (1):
- Hospital Regional Universitario de Málaga, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset contains highly sensitive genomic, transcriptomic, and immunological data from pediatric participants. Data cannot be sufficiently anonymized to ensure participant privacy under GDPR regulations. Only aggregated results will be made publicly available.